CLINICAL TRIAL: NCT02176772
Title: The Effects of Tuberculosis on Dietary Iron Absorption and Systemic Iron Utilization: a Double Stable Isotope Study in Bagamoyo, Tanzania
Brief Title: Iron Absorption and Utilization During Tuberculosis and After Treatment
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Fe_TB_Study_TZ
Record Dates: First submitted 2014-06-23; First posted 2014-06-27 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tuberculosis, no HIV and severe anemia
  Interventions: Other: Stable iron isotopes, non-drug intervention

INTERVENTIONS:
Other: Stable iron isotopes, non-drug intervention

SUMMARY:
Background: The disease burden of tuberculosis (TB), second only to HIV/AIDS among infectious diseases, is a major public health problem in developing countries. Accumulating evidence suggests that iron status is a primary determinant of TB progression. Anaemia is prevalent in patients with TB, particularly in sub-Saharan Africa, and associated with increased mortality. Anaemia in TB may be due to inflammation, dietary iron deficiency, or both, and distinguishing among these aetiologies is difficult. Iron supplementation is commonly used to treat anaemia in TB patients, but may be unnecessary if inflammation is the cause. Body iron sequestered by TB inflammation can be mobilized during treatment and used to correct the anaemia. Moreover, supplemental iron may be retained within macrophages, potentially increasing susceptibility to TB and leading to a poorer clinical outcome. Thus, better understanding of iron metabolism during TB and the aetiology of TB-related anaemia would clarify the potential role of iron in pathogenesis and optimal management of the disease.

The investigators hypothesize that: a) TB will increase circulating hepcidin and thereby impair dietary iron absorption and systemic utilization of iron, resulting in iron sequestration and anaemia; b) TB treatment and resolution of inflammation over 6 months will decrease circulating hepcidin, correcting these impairments and improving iron status and hemoglobin; c) the majority of iron utilized to replenish hemoglobin during recovery from TB will come from mobilization of sequestered iron stores rather than from iron absorption.

Objectives: Use iron stable isotopes to characterize iron balance over six months of TB treatment, and specifically to: a) quantify oral and intravenous iron incorporation (oral absorption and systemic iron utilization) at three time points during TB treatment (acute disease, after the intensive treatment phase and at completion of the continuation treatment phase); and b) determine the effect of treatment on iron mobilization from stores to replenish hemoglobin.

Methods/Subjects: Using a triple stable-isotope technique, iron absorption from labelled test meals (57Fe) and systemic iron utilization after labelled intravenous doses (54Fe, 58Fe) will be determined in 18 Tanzanian subjects with newly diagnosed pulmonary TB. The subjects will be studied at three time points (i) the day after TB diagnosis while infected, (ii) after 8 weeks of intensive phase treatment, and (iii) after another 16 weeks of continuation phase treatment. Iron status, hemoglobin, hepcidin and inflammation indexes will be measured at each time point. Isotope enrichment during the two treatment phases will be measured to estimate the relative rates of iron absorption and mobilization from stores during the intensive and continuation phases to determine the relative contributions of iron absorption and iron mobilization from stores during TB treatment and recovery.

Outcome: These studies will provide important new insights into the aetiology of anaemia and iron metabolism in TB patients. The results will provide essential data for evidence-based recommendations on the timing, administration route and efficacy of iron therapy in patients with TB, making possible, a safer and more effective treatment of anaemia in TB while decreasing morbidity and mortality from the disease.

ELIGIBILITY:
Inclusion Criteria:

* Females and males 18-45 years of age
* Sputum smear-positive, and confirmed by polymerase chain reaction and culture
* Obtained informed consent

Exclusion Criteria:

* Pregnancy or Lactating (assessed by pregnancy test)
* Body weight <40 kg
* Severe anaemia (Hb <70 g/L)
* HIV positive (assessed by HIV test)
* Positive rapid malaria antigen test
* Intake of mineral/vitamin supplements 2 weeks before and during the study
* Diagnosed metabolic or gastrointestinal disorders, eating disorders or food allergy
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 6 months
* Subject who cannot be expected to comply with study protocol (e.g. non-residents to the Bagamoyo Coast region, or subjects who plan to travel or move)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18 tuberculosis cases recruited at the Bagamoyo District Hospital and surrounding TB diagnostic centres.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in iron absorption of stable isotope tracers at week 8 | baseline, 8 weeks
  Stable iron isotopes will be orally administered under standardized conditions and close supervision. Iron absorption will be calculated from the shift in the normal isotopic abundance in red blood cells; 8 weeks = end of first treatment phase
Change from baseline in iron incorporation of stable isotope tracers at week 8 | baseline, 8 weeks
  Stable iron isotopes will be infused under standardized conditions and close supervision. Iron incorporation will be calculated from the shift in the normal isotopic abundance in red blood cells; 8 weeks = end of first treatment phase.
Change from baseline in iron absorption of stable isotope tracers at week 24 | baseline, 24 weeks
  Stable iron isotopes will be orally administered under standardized conditions and close supervision. Iron absorption will be calculated from the shift in the normal isotopic abundance in red blood cells; 24 weeks = end of second treatment phase
Change from baseline in iron incorporation of stable isotope tracers at week 24 | baseline, 24 weeks
  Stable iron isotopes will be infused under standardized conditions and close supervision. Iron incorporation will be calculated from the shift in the normal isotopic abundance in red blood cells; 24 weeks = end of second treatment phase.

SECONDARY OUTCOMES:
Change from baseline in serum hepcidin at week 2 | baseline, 2 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 4 | baseline, 4 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 6 | baseline, 6 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 8 | baseline, 8 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 10 | baseline, 10 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 12 | baseline, 12 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 14 | baseline, 14 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 16 | baseline, 16 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 18 | baseline, 18 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 20 | baseline, 20 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 22 | baseline, 22 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 24 | baseline, 24 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.
Change from baseline in serum hepcidin at week 26 | baseline, 26 weeks
  As a determinant of iron metabolism, serum hepcidin will be measured several times during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Tb-clinic, Bagamoyo Research and Training Centre, Bagamoyo, Coast Region, Tanzania

REFERENCES:
- [Derived] Cercamondi CI, Stoffel NU, Moretti D, Zoller T, Swinkels DW, Zeder C, Mhimibra F, Hella J, Fenner L, Zimmermann MB. Iron homeostasis during anemia of inflammation: a prospective study of patients with tuberculosis. Blood. 2021 Oct 14;138(15):1293-1303. doi: 10.1182/blood.2020010562. PMID 33876222